CLINICAL TRIAL: NCT03888989
Title: Response to Influenza Vaccine During Pregnancy
Acronym: FLU-PG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment was not complete given logistical concerns that arose during the COVID-19 pandemic
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 50163; 5U19AI057229-15 (NIH)
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Influenza
Keywords: Influenza; Pregnancy; Quadrivalent inactivated influenza vaccine (IIV).
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Phase (Other): Participants will be given the current year's quadrivalent inactivated influenza vaccine (IIV)
  Interventions: Biological: Quadrivalent inactivated influenza vaccine (IIV)

INTERVENTIONS:
Biological: Quadrivalent inactivated influenza vaccine (IIV) — Quadrivalent inactivated influenza vaccine (IIV), Intramuscular Injection

SUMMARY:
This is one project of a larger ongoing study related to the immune system's response to the flu virus. This study is designed to investigate the immune response to vaccination in pregnancy.

DETAILED DESCRIPTION:
This is a Phase I mechanistic study of licensed influenza vaccines with up to 50 pregnant female volunteers, 18-49 years of age. Investigator intends to collect blood from pregnant women and then from the same women a year later when they are not pregnant after routine seasonal influenza vaccination. By studying the blood of immunized pregnant women and in these same women after pregnancy, the investigator will gain a better understanding of the immune response to vaccination in pregnancy and after pregnancy.

Each volunteer will participate for approximately 4 weeks including enrollment, vaccination, and completion of sample collection in 2 consecutive flu seasons. The Study has a total of 6 visits over 2 Flu seasons.

Study procedures:

Year One:

First Visit: Procedures during this visit are: Informed consent process, enrollment, study assessments, 20 ml blood draw, and vaccination.

2nd and 3rd visits: 20 ml blood will be obtained

Year Two:

First Visit: Study assessments, 20 ml blood draw, and vaccination. 2nd and 3rd visits: 20 ml blood will be obtained

ELIGIBILITY:
Inclusion Criteria:

1. 18-49-year-old pregnant woman
2. Willing and able to complete the informed consent process
3. Availability for follow-up for the planned duration of the study with the expected delivery date more than 28 days after vaccination
4. Acceptable medical history by review of inclusion/exclusion criteria

Exclusion Criteria:

1. Prior off-study vaccination with seasonal influenza vaccine within three months of study vaccination
2. Life-threatening reactions to previous influenza vaccinations
3. Allergy to egg or egg products or to vaccine components including gentamicin, gelatin, or arginine.
4. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
5. History of immunodeficiency (including HIV infection)
6. Known or suspected impairment of immunologic function; may include significant liver disease, diabetes mellitus treated with insulin or moderate to severe renal disease
7. Chronic Hepatitis B or C.
8. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
9. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
10. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator might jeopardize volunteer safety or compliance with the protocol.
11. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
12. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox will be reviewed by investigators to determine if study participation would affect the volunteer's safety or compliance with the protocol.
13. Receipt of blood or blood products within the past 6 months or planned used during the study.
14. A medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
15. Receipt of an inactivated vaccine 14 days prior to study enrollment, or planned vaccinations prior to completion of last annual study visit (~ 28 days after study vaccination)
16. Receipt of a live, attenuated vaccine within 60 days prior to enrollment of planned vaccination prior to completion of last study visit (~ 28 days after study enrollment)
17. Need for allergy immunization (that cannot be postponed) until after the last study visit.
18. History of Guillain-Barre# syndrome
19. Use of investigational agents within 30 days prior to enrollment or planned use during the study.
20. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment or donation of platelets within 2 weeks of enrollment or planned donation prior to completion of the last visit.
21. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Females
Enrollment: 2 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Grant, Principal Investigator — Assistant Professor of Medicine (Infectious Diseases)
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Phase
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Inactivated Influenza Vaccine: Participants received the annual IIV
Arm/Group | Inactivated Influenza Vaccine
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 29 [25 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Plasma HAI Titer at Day 7 (Year 1)
Description: HAI titer measures immune response to influenza vaccination. An HAI titer is a hemoglobin assay that correlates to protection from influenza infection; an HAI titer of 40 or greater is considered to be protective.
Time Frame: Day 7 (after year 1 vaccine administration)
Population: Data were not collected for this outcome measure.
Groups:
- Participants Who Received IIV: Participants who received IIV
Arm/Group | Participants Who Received IIV
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Related Adverse Events (Year 1)
Description: AEs related to IIV
Time Frame: Baseline to Day 28 post year 1 vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received IIV
Number analyzed (Participants) | 2
Participants | 0

3. Primary Outcome: Number of Participants With Related Adverse Events (Year 2)
Description: AEs to IIV
Time Frame: Baseline to Day 28 post year 2 vaccine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received IIV
Number analyzed (Participants) | 2
Participants | 0

4. Primary Outcome: Plasma HAI Titer at Day 7 (Year 2)
Description: as for outcome 1
Time Frame: Day 7 (Year 2)
Population: Data were not collected for this outcome measure.
Arm/Group | Participants Who Received IIV
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to Day 28 post year 2 vaccine administration
Arm/Group | Study Phase
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The Covid-19 pandemic led to early termination and a very small numbers of subjects recruited and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03888989/Prot_000.pdf
  • Informed Consent Form (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT03888989/ICF_001.pdf